CLINICAL TRIAL: NCT07189026
Title: Prevalence and Clinical Impact of Airway Opening Pressure in Post-Cardiac Surgery Patients: A Prospective Observational Study
Brief Title: Prevalence and Clinical Impact of Airway Opening Pressure in Post-Cardiac Surgery Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2026-4399
Record Dates: First submitted 2025-08-27; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery; Mechanical Ventilation After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post operative cardiac surgery (Other)
  Interventions: Diagnostic Test: Airway opening pressure

INTERVENTIONS:
Diagnostic Test: Airway opening pressure — Airway opening pressure will be measured within one hour of intensive care unit admission (using a standardized low-flow insufflation maneuver flow 5-6 LPM). The inflection point on the pressure-time or pressure-volume waveform- depending on ventilator model-will define the airway opening pressure.

SUMMARY:
Airway opening pressure is a key parameter in assessing respiratory mechanics. Current practice primarily relies on indirect assessments of lung mechanics, but growing evidence suggests that direct airway opening pressure measurement could enhance individualized ventilatory strategies. Significant airway opening pressure suggests incomplete alveolar recruitment at end-expiration, which may contribute to ventilation-perfusion mismatch, increased respiratory effort, and postoperative pulmonary complications such as atelectasis and impaired gas exchange. Determining the prevalence and clinical relevance of significant airway opening pressure in post-cardiac surgery patients could contribute to more personalized respiratory strategies and improve postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Undergoing elective coronary artery bypass grafting (CABG) or valve surgery, or combined procedures with expected postoperative mechanical ventilation

Exclusion Criteria:

- Patient receiving invasive mechanical ventilation prior to surgery

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of significant airway opening pressure | up to 1 hour after intensive care admission
  airway opening pressure ≥ 5 cmH₂O

SECONDARY OUTCOMES:
Airway opening pressure prevalence based on body mass index | up to 1 hour
  Airway opening pressure prevalence base on Obesity status (body mass index ≥30 vs. <30 kg/m²)
Airway opening pressure prevalence based on cardiopulmonary bypass duration | up to 1 hour
  Airway opening pressure prevalence based on cardiopulmonary bypass duration (minutes)
Airway opening pressure prevalence based on left ventricular dysfunction | up to 1 hour
  Airway opening pressure prevalence based on left ventricular dysfunction (Ieft ventricular ejection fraction < 50 percent vs > 50 percent)
Airway opening pressure prevalence based on inotropic support | up to 1 hour
  Airway opening pressure prevalence based on use of amines (< 0.1 mcg/kg/min or norepinephrine equivalent vs > 0.1 mcg/kg/min or norepinephrine equivalent)
Airway opening pressure prevalence based on age | up to 1 hour
  Airway opening pressure prevalence base on age
Airway opening pressure prevalence based on intraoperative fluid balance | up to 1 hour
  Airway opening pressure prevalence base on intraoperative fluid balance
Feasibility of airway opening pressure measurement | up to 1 hour
  proportion of patients in whom the maneuver is successfully completed
Positive end expiratory pressure level | up to 1 hour
  Number of times Positive end expiratory pressure is set greater than measured airway opening pressure
Extubation | Day7
  Correlation between airway opening pressure and time to extubation
Patient position | up to 1 hour
  Comparison of airway opening pressure values in flat versus semi-recumbent (30-degree) positions
Hemodynamic tolerance base on blood pressure drop | up to 15 minutes
  Evaluation of hemodynamic tolerance based on arterial pressure during positive end-expiratory pressure adjustment (if inotropic agents are required, an increase of more than 0.05 mcg/kg/min in norepinephrine equivalent is considered significant)
Hemodynamic tolerance base on pulse oxygen saturation drop | up to 15 minutes
  Evaluation of hemodynamic tolerance based on pulse oxygen saturation. A decrease in pulse oxygen saturation of 5 percent from baseline or more is considered significant.
Non-interruptive airway opening pressure measurement method | up to 1 hour
  The novel non-interruptive airway opening pressure measurement method will be validated

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No